CLINICAL TRIAL: NCT04500418
Title: Charité Trial of Cenicriviroc (CVC) Treatment for COVID-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite multiple efforts, no further patient could be enrolled since 03/05/2021. A continuation of the study is therefore no longer justified
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Frank Tacke, Prof. Dr. med., PhD, MHBA, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVC for COVID-19; 2020-001493-29 (EudraCT Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: COVID-19; Cenicriviroc; CVC; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — cenicriviroc

STUDY DESIGN:
Intervention Model Description: A monocentric, randomized, double-blind, placebo-controlled trial.
  Randomization will be stratified by:
  * Presence of baseline score of "3" on 7-point ordinal scale versus presence of baseline score of "4" or "5" on seven-point ordinal scale
  * Presence of one or more of the following comorbidities: Diabetes mellitus, Obesity (BMI >30kg/m2), COPD or Asthma, Heart failure (NYHA Class I or II)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cenicriviroc (CVC) (Active Comparator): Approximately 122 patients. Day 1: CVC 450 mg (300 mg AM; 150 mg PM; if patients receive their first dose on Day 1 past 2 PM, then their evening dose will be 300 mg and their next dose will be the following AM.) Days 2-28: CVC BID 150 mg (AM/PM). Every dose should be taken with food (within 30 min).
  Interventions: Drug: Cenicriviroc (CVC)
- Placebo (Placebo Comparator): Approximately 61 patients. A matching placebo will be given to the patients in the Placebo group at an equal volume and at the same schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenicriviroc (CVC) — Treatment with Cenicriviroc tablets of 150mg. (450g/300g on day 1 and 300mg/d on days 2-28).
  Other Names: Cenicriviroc Mesylate
  Arms: Cenicriviroc (CVC)
Drug: Placebo — Optically identical pills without CVC.
  Arms: Placebo

SUMMARY:
The aim of this study is to test Cenicriviroc (CVC) as a means to reduce the severity of the lung disease COVID-19 caused by an infection with SARS-CoV-2. The safety of CVC, when administered to COVID-19 patients, will also be assessed. Furthermore, the clinical trial aims to answer the question of whether patients with pre-existing conditions, who have an increased risk of severe COVID-19 progression, benefit more and particularly from CVC. CVC is an orally available dual inhibitor of the chemokine receptors CCR2 and CCR5, which is expected to reduce (hyper-) inflammation in COVID-19.

The main goal of the study is to determine whether CVC helps increase the number of patients who are symptom-free and not hospitalized after 14 days compared to a placebo. Approximately 66.7% of the patients enrolled in the study will receive CVC and 33.3% will get an optically identical pill (placebo).

Subjects will be assessed daily while hospitalized. Discharged patients will be asked to attend study visits at Days 8, 15, 22, and 29 and 85. All subjects will undergo a series of clinical, safety, and laboratory assessments. Blood samples and oropharyngeal (OP) swabs will be obtained on Day 1; 3, 5 (while hospitalized); and Day 8, 15 and 29 (if able to return to clinic or still hospitalized). The presence of anti-SARS-CoV-2 antibodies will be determined on Days 29 and 85.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent prior to initiation of any study procedures. Understands and agrees to comply with planned study procedures.
* Male or non-pregnant female adult ≥18 years of age at time of enrolment.
* Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR and fulfils the case criteria of COVID-19 (One or more of the following must be met in lieu of a positive PCR test: fever [defined as a temperature ≥ 100.0°F / 37.8°C documented within 24 hr. of randomization] , absolute and relative lymphopenia and leukopenia, new typical infiltrates in x-ray of the chest or chest CT scan [only if obtained for clinical reasons; not required by study], no improvement on antibiotics).
* Scoring a "3" or "4" (or "5", at the Investigator's discretion) on the 7-Point Ordinal Scale (see Outcome Measures) at enrolment. Note, if scoring a "2" at screening, inclusion will be met if the patient is in the process of being hospitalized or admitted to an inpatient setting. Such a patient would be assigned a "3" at enrolment for Baseline assessment purposes.
* No participation in other clinical trials according to the German Medicines Act (AMG) (3 months before) at the time of this trial.

Exclusion Criteria:

* ALT/AST > 5 times the upper limit of normal.
* Patients with severe hepatic impairment (defined as liver cirrhosis Child stage B or C)
* Stage 4 chronic kidney disease or requiring dialysis (i.e. eGFR < 30 ml/min)
* Advanced cardiac (eg, severe heart failure [NYHA III-IV]) or pulmonary diseases which, in the Investigator's judgment, would not make participation appropriate.
* Pregnancy or breast feeding.
* Anticipated transfer to another hospital which is not a study site within 72 hours.
* Known allergy or hypersensitivity to CVC or its components.
* Use of medications that are contraindicated with CVC and that could not be replaced or stopped during the trial period
* Administration of specified drugs which interfere with the metabolism of CVC.
* Patients immediately or imminently requiring mechanical ventilation.
* Patients unwilling to consent to saving and propagation of pseudonymised medical data for study reasons.
* Subjects who are legally detained in an official institution.
* Subjects that are unsuitable to understand or to comply with the study requirements in the opinion of the investigator.
* Subjects who may be dependent on the sponsor, the investigator or the trial sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Subject´s Responder status (score on the 7-point ordinal scale on Day 15) | 14 days after enrollment (Day 15)
  The Primary Endpoint will be the subject's responder status defined by achieving a score of "1" or "2" (discharged from hospital e.g.) on Day 15 on the following 7-point scale:
  1. Not hospitalized, no limitations on activities;
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high-flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO (Extracorporeal membrane oxygenation);
  7. Death.

SECONDARY OUTCOMES:
Evaluation of change in clinical condition based on the 7-point ordinal scale | day of enrollment and 15 days after enrollment
  7-point ordinal scale to be assessed on Day 15 (and Day 1 for baseline comparison), analyses of
  * ordinal change of 2 or more, compared with baseline
  * ordinal change of 1 or more, compared with baseline
Evaluation of change in clinical condition based on the 7-point ordinal scale and Responder Status | day of enrollment, 8 days, 22 days and 29 days after enrollment
  7-point ordinal scale assessed on: Days 8, 22, 29 (and Day 1 for baseline comparison), analyses of:
  * Responder status (achieving a score of a "1" or a "2")
  * ordinal change of 2 or more, compared with baseline
  * ordinal change of 1 or more, compared with baseline
Hospital resource utilization comparison | 29 days after enrollment, 85 days after enrollment
  Analysis of:
  * Length of time spent in the ICU (days)
  * Length of time spent in the hospital (days)
  * Days alive and out of hospital through Day 29
  * Days free of endotracheal tube-based ventilation through Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tacke, Prof. Dr.med., Principal Investigator — Charité University, Berlin, Germany
Locations (1):
- Medical Department of Hepatology and Gastroenterology, Charité University Medicine, Campus Virchow Klinikum (CVK) and Campus Charité Mitte (CCM), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this moment. (08/2020)